CLINICAL TRIAL: NCT04344808
Title: Accuracy and Patient-Reported Outcome Measures (PROMs) of a Dynamic Navigation System in Implantology: A Randomized Controlled Trial
Brief Title: Dynamic Navigation System in Implantology
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Barcelona (Other)
Responsible Party: Principal Investigator, Rui Figueiredo, Associate Professor. PhD, MD, DDS, University of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NavigationSystem
Record Dates: First submitted 2020-03-30; First posted 2020-04-14 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Surgery, Computer-Assisted; Dental Implants
Keywords: Surgery, Computer-Assisted; Dental Implants; Navigation system; Dynamic computer-assisted surgery; Implantology

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patient will be unaware of which group since during the surgical procedure patient eyes' will be covered.
  Outcome assessor won't take part of the clinical process and will be blinded regarding which group is allocated each patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Navigation group (Experimental): Dental implants will be placed using a dynamic computer assisted surgery system
  Interventions: Device: Dynamic navigation system
- Freehand group (Active Comparator): Dental implants will be place without any guidance. Only virtually planning the ideal position on a 3D image (Cone beam computed tomography)
  Interventions: Device: Freehand implant placement

INTERVENTIONS:
Device: Dynamic navigation system — The navigation system allows clinicians, using a specific software, to visualize the position of the surgical drill (tip location and shaft axis direction) on the reconstructed 3D image of the pre-acquired CBCT. The software guides the surgeon, in real-time, to the preoperative planned position.
  Other Names: Dynamic computer assisted surgery
  Arms: Navigation group
Device: Freehand implant placement — Dental implants will be placed without any guidance once a virtually planning of the ideal position on the CBCT is done
  Other Names: Non-guided implant placement
  Arms: Freehand group

SUMMARY:
This study consists in a randomized controlled trial which objective is to assess the accuracy of a dynamic navigation system in dental implant placement in partially edentulous patients compared with the conventional freehand method.

DETAILED DESCRIPTION:
This is a prospective randomized clinical trial.

Each patient enrolled in this trial will be randomly allocated to one group ( Navigation group or Freehand groups). Preoperative virtual planification of dental implants on a pre-acquired cone beam computed tomography (CBCT) will be performed for each patient using the same system.

During the surgical phase, depending on which group is allocated the patient one surgical approach or other will be used. Then after the surgical procedure a PROMs questionnaire will be asked to the patients.

Finally a postoperative CBCT will be performed and overlapped with the preoperative CBCT (with the implants planification) and implant position deviations between the planned and final position will be measured.

The study devices are CE- (Conformité Européenne, meaning European Conformity) marked products and used within their intended use.

ELIGIBILITY:
Inclusion Criteria:

* Partially edentulous patients that requires at least the placement of one dental implant
* Healthy patients ASA I and II (American Society of Anesthesiologists classification)
* Over 18 years old patients

Exclusion Criteria:

* Totally edentulous patients
* Systemic or local conditions that contraindicates dental implant surgery
* Patients with less than 3 teeth in the jaw.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Angular deviation | 3 months post operative
  angular deviation between the virtual planed position of the implant and the final implant position. Measured in degrees
Platform 3D deviation | 3 months post operative
  global deviation at the platform of the dental implant between the virtual planned position and the final position of the dental implant measured in the 3 axes of the space (3D deviation). Measured in millimeters (mm).
Apex 3D deviation | 3 months post operative
  global deviation at the apex of the dental implant between the virtual planned position and the final position of the dental implant measured in the 3 axes of the space (3D deviation). Measured in millimeters (mm).
Platform 2D deviation | 3 months post operative
  Lateral deviation at the platform of the dental implant between the virtual planned position and the final position of the dental implant measured in 2 axes of the space (x and y, 2D deviation). Measured in millimeters (mm).
Apex depth deviation | 3 months post operative
  Depth deviation of the apex of the dental implant between the virtual planned position and the final position of the dental implant in the Z-axis. Measured in millimeters (mm).

SECONDARY OUTCOMES:
Patient-reported outcome measures (PROMs) questionnaire | One week post operative.
  Patients perception of their functional well-being and health status during the dental implant treatment with a navigation system. We will use OHIP-14 (Oral Health Impact Profile) questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Adrià Jorba-García, Principal Investigator — University of Barcelona; Rui Figueiredo, Study Director — University of Barcelona; Eduard Valmaseda-Castellón, Study Chair — University of Barcelona; Octavi Camps-Font, Study Chair — University of Barcelona; Javier Bara-Casaus, Study Chair — University of Barcelona
Locations (1):
- Universitat de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vercruyssen M, Fortin T, Widmann G, Jacobs R, Quirynen M. Different techniques of static/dynamic guided implant surgery: modalities and indications. Periodontol 2000. 2014 Oct;66(1):214-27. doi: 10.1111/prd.12056. PMID 25123770
- [Background] Aydemir CA, Arisan V. Accuracy of dental implant placement via dynamic navigation or the freehand method: A split-mouth randomized controlled clinical trial. Clin Oral Implants Res. 2020 Mar;31(3):255-263. doi: 10.1111/clr.13563. Epub 2019 Dec 29. PMID 31829457
- [Background] D'haese J, Ackhurst J, Wismeijer D, De Bruyn H, Tahmaseb A. Current state of the art of computer-guided implant surgery. Periodontol 2000. 2017 Feb;73(1):121-133. doi: 10.1111/prd.12175. PMID 28000275
- [Background] Jorba-Garcia A, Figueiredo R, Gonzalez-Barnadas A, Camps-Font O, Valmaseda-Castellon E. Accuracy and the role of experience in dynamic computer guided dental implant surgery: An in-vitro study. Med Oral Patol Oral Cir Bucal. 2019 Jan 1;24(1):e76-e83. doi: 10.4317/medoral.22785. PMID 30573712
- [Background] Block MS, Emery RW. Static or Dynamic Navigation for Implant Placement-Choosing the Method of Guidance. J Oral Maxillofac Surg. 2016 Feb;74(2):269-77. doi: 10.1016/j.joms.2015.09.022. Epub 2015 Sep 30. PMID 26452429
- [Background] Emery RW, Merritt SA, Lank K, Gibbs JD. Accuracy of Dynamic Navigation for Dental Implant Placement-Model-Based Evaluation. J Oral Implantol. 2016 Oct;42(5):399-405. doi: 10.1563/aaid-joi-D-16-00025. Epub 2016 Jun 6. PMID 27267658
- [Background] Jung RE, Schneider D, Ganeles J, Wismeijer D, Zwahlen M, Hammerle CH, Tahmaseb A. Computer technology applications in surgical implant dentistry: a systematic review. Int J Oral Maxillofac Implants. 2009;24 Suppl:92-109. PMID 19885437